CLINICAL TRIAL: NCT02049853
Title: A Prospective Randomized Study of Coordinated Diagnostic Pathways and Treatment Algorithms for Patients With Acute Dyspnea Including Point-of-care Testing of a Cardiac Biomarker by the Emergency Medical Service Team
Brief Title: The Triple A Initiative Study ("Aktionsbündnis Akute Atemnot")
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment numbers lower than expected
Sponsor: Prof. Dr. Michael Christ (Other)
Collaborators: Jena University Hospital (Other); City Hospital Fürth (Other); Roche Pharma AG (Industry); Bayrisches Rotes Kreuz Fuerth (Unknown); Johanniter Unfall Hilfe Nürnberg (Unknown); DRK-Kreisverbandes Jena-Eisenberg-Stadtroda e.V. (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Dr. Michael Christ, Prof. Dr. med. Michael Christ, Klinikum Nürnberg
Organization: Klinikum Nürnberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TripleA01
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Dyspnea; Heart Failure
Keywords: acute dyspnea; heart failure; diagnostics; POCT analysis; preclinical area
MeSH Terms: conditions — Dyspnea; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- default group (No Intervention): Patients with the randomization result "default group" receive standard diagnostics
- POCT group (Active Comparator): patients with the randomization result "POCT group" receive a NTproBNP measurement with point of care device "Cobash232" in the ambulance vehicle
  Interventions: Device: NTproBNP measurement with point of care device "Cobash232" in the POCT group

INTERVENTIONS:
Device: NTproBNP measurement with point of care device "Cobash232" in the POCT group
  Arms: POCT group

SUMMARY:
Acute dyspnea is a common chief complaint of patients presenting to the emergency department. Patients with acute dyspnea display a high mortality rate. In-hospital mortality is as high as 10% during hospitalization and up to 30% within 6 months of follow-up. The Triple A Initiative Study is designed to improve the coordination of care for patients with acute dyspnea alerting the Emergency Medical Service (EMS). We hypothesize that the coordination of care starting at the EMS level including point-of-care testing of the cardiac biomarker NTproBNP will support preclinical and clinical diagnostic clarification. Treatment deriving from earlier diagnostic clarification will reduce length of stay in the hospital, treatment costs and improve patient's outcome.

DETAILED DESCRIPTION:
The aim of this prospective, randomized study is to evaluate the effects of point-of-care testing of NT-proBNP in patients presenting with acute dyspnea to the Emergency Medical Service (EMS).Patients will be enrolled in the Emergency Medical Services of participating German hospitals (Klinikum Nürnberg, Klinikum Fürth, Universitätsklinikum Jena). To be enrolled in the study, each patient must meet all of the following inclusion criteria and none of the exclusion criteria.

Patients with acute dyspnea randomized to the POCT group will get a NT-proBNP-POCT measurement in the EMS. The emergency physician of the EMS will decide to apply predefined treatment strategies according to the resulting working hypothesis. Patients with acute dyspnea randomized to the standard care group will NOT get NT-proBNP measurement at the scene. The emergency physician of the ED will construct the working hypothesis following current treatment recommendations. The major focus of the study is to initiate treatment of heart failure as early as possible.

ELIGIBILITY:
Inclusion Criteria:

* acute dyspnea (NYHA II-IV)
* age >= 18 years
* informed consent

Exclusion Criteria:

* cardiopulmonary resuscitation < 7 days
* cardiogenic shock, STEMI, respiratory failure, or other clinical conditions that require immediate intensive care admission or angioplasty
* systolic blood pressure lower than 100 mmHg at first contact/presentation
* ventricular tachycardia
* severe aortic stenosis
* advanced neoplasm (e.g. lung cancer, hematologic neoplasm, etc.)
* chronic kidney disease requiring hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2013-06; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Days alive and out of hospital within 30 days | 30 days

SECONDARY OUTCOMES:
Cost-effectiveness analysis evaluating both costs and effects of alternative therapies (NT-proBNP vs. control group) at day 30, 90 and 180 days | 60 months
Diagnostic accuracy of chest ultrasound to detect patients with acute heart failure | 1 month
In-hospital length of stay during follow-up of 30 and 90 days | 3 months
Improvement of symptoms (dyspnea) 24h, 48h, 72h hours after admission | 1 month
Need for ICU admission during initial hospitalization | 6 months
B-type natriuretic peptide level and calculated glomerular filtration rate at discharge | 6 months
Patients functional status at 30, 90 and 180 days (Barthel Index) | 6 months
Mortality at 30, 90 and 180 days | 6 months
Total treatment costs at 30, 90 and 180 days | 6 months
Days alive and out of hospital at 90 and 180 days | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Christ, Prof., Principal Investigator — Klinikum Nürnberg
Locations (6):
- Germany (6):
  - Klinikum Nürnberg, Nuremberg, Bavaria
  - Bayrisches Rotes Kreuz, Fürth
  - Klinikum Fürth, Emergency Department, Fürth
  - Universitätsklinikum Jena, Department of Anesthesiology and Intensive Care Medicine, Jena
  - DRK-Kreisverbandes Jena-Eisenberg-Stadtroda e.V., Jena
  - Johanniter-Unfall-Hilfe, Nuremberg